CLINICAL TRIAL: NCT00346476
Title: A Study of the Effects of Antiretroviral Therapy on Rates and Transmission of Tuberculosis
Brief Title: Characteristics and Prevalence of Tuberculosis and HIV in Masiphumelele Township, Cape Town, South Africa
Status: Completed | Type: Observational
Sponsor: CIPRA SA (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Comprehensive International Program of Research on AIDS (Other)
Responsible Party: James McIntyre, CIPRA SA
Other Study IDs: CIPRA-SA Project 3B; U19AI053217 (NIH)
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections; Tuberculosis
Keywords: TB; Transmission; Genetic Diversity; Genetic Testing; RFLP
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Individuals in the Masiphumelele Township of Cape Town, South Africa, who have been potentially exposed to TB and/or HIV

SUMMARY:
The purpose of this study is to determine the number of people infected with tuberculosis (TB) in the Masiphumelele Township of Cape Town, South Africa, a community with high rates of TB and HIV. This study will also examine the genetics of TB and the relationships among active TB infection, new HIV infections, and HIV disease progression.

DETAILED DESCRIPTION:
TB is the most common opportunistic infection and the single most common cause of death in HIV infected people in Africa today. Latent TB infection has been known to revert to active TB following new infection in HIV infected people; also, TB has been shown to accelerate the progression of HIV disease. These epidemiologic relationships between TB and HIV and the high prevalence of these diseases in sub-Saharan Africa make studying TB and HIV infected populations in this region of the world important. The Masiphumelele Township of Cape Town, South Africa, with its high rates of TB and HIV, is representative of many poor communities in Africa. The purpose of this study is to observe people from the Masiphumelele Township over a 5-year period to assess the prevalence of TB and HIV infections in a random sample of people and the clinical and genetic characteristics of active TB infection.

This study has two parts: a random cross-sectional survey and a clinical and genetic assessment of TB patients. Participants in the random survey will only be involved with the study for a maximum of 2 days. The purpose of the first part of the study is to compare the prevalence of active TB and the prevalence of HIV infection in a random sample of people from the Masiphumelele Township. In this part of the study, children and adults will be randomly selected from the township population to determine the prevalence of active TB and the prevalence of HIV infection in this group of people. Fieldworkers will identify eligible participants in the township and will ask them to visit the clinic that day or the next. At the clinic, participants will be asked to complete a demographics and TB history questionnaire and provide a saliva sample for anonymous HIV testing. A sputum sample will be collected from each participant with a nebulizer; each participant will also be given a sputum sample bottle and will be asked to collect an early morning sputum sample on the next day that will be returned to the clinic.

The second part of the study will enroll TB patients. Participants in this part of this study will be followed for the course of their TB treatment for at least 6 months. The purpose of the second part of the study is to assess changes through time of the clustering and transmission of TB among HIV infected and uninfected people in the Masiphumelele Township. This assessment will include examining the diversity of TB strains in this population and determining the relationship between recurrent cases of TB and HIV infection. All sputum samples indicating TB infections that were previously collected from participants will undergo genetic testing by restriction fragment length polymorphism (RFLP) analysis. Participants will be asked to complete a demographics and TB history questionnaire and provide a saliva sample for anonymous HIV testing. Participants will also be interviewed about treatment they have received for TB, their responses to this treatment, and whether they are currently on highly active antiretroviral therapy (HAART) for the treatment of HIV infection.

Participants who are found to be infected with TB during the first part of the study will be offered TB treatment through the clinic and will be invited to participate in the second part of this study. Participants who are found to be infected with HIV during the study will be referred to further treatment and evaluation.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Willing to comply with study requirements
* Parent or guardian willing to provide informed consent, if applicable

Inclusion Criteria for Participants in First Part of the Study:

* Live in Masiphumelele Township, Cape Town, South Africa for at least 1 week

Inclusion Criteria for Participants in Second Part of the Study:

* Live in Masiphumelele Township, Cape Town, South Africa
* Registered TB patient at the study site

Exclusion Criteria for All Participants:

* Currently incarcerated

Exclusion Criteria for Participants in Second Part of the Study:

* No Mycobacterium tuberculosis specimen obtained from the participant for genetic analysis

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV and TB infected and uninfected individuals
Sampling Method: Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2006-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Gail Bekker, MBChB, FCP, PhD, Study Chair — Department of Medicine, University of Cape Town; James McIntyre, MBChB, MRCOG, Principal Investigator — University of the Witwatersrand, Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital
Locations (2):
- South Africa (2):
  - Desmond Tutu HIV Centre Department of Medicine, Cape Town, Western Cape
  - Desmond Tutu HIV Centre Department of Medicine, Cape Town

REFERENCES:
- [Background] Aaron L, Saadoun D, Calatroni I, Launay O, Memain N, Vincent V, Marchal G, Dupont B, Bouchaud O, Valeyre D, Lortholary O. Tuberculosis in HIV-infected patients: a comprehensive review. Clin Microbiol Infect. 2004 May;10(5):388-98. doi: 10.1111/j.1469-0691.2004.00758.x. PMID 15113314
- [Background] Badri M, Ehrlich R, Wood R, Pulerwitz T, Maartens G. Association between tuberculosis and HIV disease progression in a high tuberculosis prevalence area. Int J Tuberc Lung Dis. 2001 Mar;5(3):225-32. PMID 11326821
- [Background] Friedland G, Harries A, Coetzee D. Implementation issues in tuberculosis/HIV program collaboration and integration: 3 case studies. J Infect Dis. 2007 Aug 15;196 Suppl 1:S114-23. doi: 10.1086/518664. PMID 17624820
- [Background] Kwara A, Flanigan TP, Carter EJ. Highly active antiretroviral therapy (HAART) in adults with tuberculosis: current status. Int J Tuberc Lung Dis. 2005 Mar;9(3):248-57. PMID 15786886
- [Background] Maher D, Harries A, Getahun H. Tuberculosis and HIV interaction in sub-Saharan Africa: impact on patients and programmes; implications for policies. Trop Med Int Health. 2005 Aug;10(8):734-42. doi: 10.1111/j.1365-3156.2005.01456.x. PMID 16045459
- [Background] Perkins MD, Cunningham J. Facing the crisis: improving the diagnosis of tuberculosis in the HIV era. J Infect Dis. 2007 Aug 15;196 Suppl 1:S15-27. doi: 10.1086/518656. PMID 17624822
- [Background] Wood R, Maartens G, Lombard CJ. Risk factors for developing tuberculosis in HIV-1-infected adults from communities with a low or very high incidence of tuberculosis. J Acquir Immune Defic Syndr. 2000 Jan 1;23(1):75-80. doi: 10.1097/00126334-200001010-00010. PMID 10708059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants
Started | 1250
Completed | 1250
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 1250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55
  Between 18 and 65 years | 1185
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 28.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 602
  Male | 648
Region of Enrollment [Number; unit: participants]
  South Africa | 1250

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Microbiologically Confirmed Tuberculosis Infection
Time Frame: At Year 5
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 1250
participants | 20

2. Secondary Outcome: Changes in Clustering and Transmission of TB Among HIV Infected and Uninfected Participants
Time Frame: Year 1 to Year 5
Reporting Status: Not Posted

3. Secondary Outcome: Changes in the Clustering and Transmission of TB Among HIV Infected and Uninfected Participants After the Introduction of HAART
Time Frame: Year 1 to Year 5
Reporting Status: Not Posted

4. Secondary Outcome: Diversity of TB Strains Among HIV Infected Participants Receiving HAART, HIV Infected Participants Not Receiving HAART, and HIV Uninfected Participants
Time Frame: Year 1 to Year 5
Reporting Status: Not Posted

5. Secondary Outcome: Number of Recurrent Cases of TB Attributable to Endogenous Reactivation Versus Exogenous Re-infection in Both HIV Infected and Uninfected Participants
Time Frame: At Year 5
Reporting Status: Not Posted

6. Primary Outcome: Number of Participants With HIV Infection
Time Frame: At Year 5
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 1250
participants | 306

ADVERSE EVENTS:
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 0/1250
Other Adverse Events (participants affected / at risk) | 0/1250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes